CLINICAL TRIAL: NCT00431509
Title: A Randomized Trial Comparing Navigated and Conventional Implantation Techniques in Knee Replacement Surgery. Influence on Operative Result, Health-Related Quality of Life, and Coordinative Abilities.
Brief Title: Trial Comparing Navigated and Conventional Implantation Techniques in Knee Replacement Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: DePuy International (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCTTKR1
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Arthroplasty; Replacement; Knee; Instrumentation
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Procedure: conventional vs. navigated total knee arthroplasty

SUMMARY:
This study is undertaken to investigate the effect of navigated knee implantation surgery on physical function, joint stiffness, pain, quality of life and coordinative abilities.

One group of patients will receive navigated knee implantation surgery, the other traditional knee implantation surgery, without use of the navigation system.

The study is designed as a randomized trial. That means that all patients who have given their consent to participate in this study will be allocated to either navigated or conventional surgery by chance.

A total of 477 patients will be included in this study and will be followed up for 12 month.

In this period all patients will be asked to fill in functional and quality of life questionnaires at baseline, 6 weeks and 3, 6 and 12 month follow-up. Coordinative abilities will be evaluated once in the time-frame 3 to 6 months postoperatively.

DETAILED DESCRIPTION:
Various risk factors influencing the success of Total Knee Arthroplasty (TKA) have been studied.

Today age, gender, primary or revision surgery, comorbidities and baseline characteristics are known to influence the health-related quality of life after TKA.

It is thought, that accurate mechanical alignment and ligament balance ensure optimal kinematic performance and wear, which in turn improves long-term outcome.

During preparation of the bone for the implantation of the knee prosthesis, numerous cuts are performed. Traditionally mechanical adjusted jigs are used to accurately align and position the instruments.

Since this alignment process is a source for deviation even in experienced surgeons, several navigation systems were developed. Using these systems, the surgeon is guided in the location of the instruments with the help of a computer.

Several studies could show that the use of such a navigation system leads to an improved execution of planned axis relations, as measured on the radiographs. However, it is not clear, whether or to what extent the improved realization of the preoperative planned axis relations results in a positive effect for the patient.

This multicenter randomized clinical trail is conducted to compare the operative results of navigated and non-navigated knee replacement surgery.

The aim of this study is to evaluate the use of a navigation system on health-related quality of life, measured as pain, stiffness, physical function, coordinative abilities, and patient satisfaction.

The hypotheses tested is that the use of the navigation system for total knee arthroplasty leads to improved health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled to receive a Total Knee Arthroplasty at the participating institutions for primary diagnosis of osteoarthritis are candidates for inclusion in the study.

Exclusion Criteria:

* A history of septic arthritis in the joint to operate
* Amputations
* Neurological deficits
* Inability to complete the questionnaires because of cognitive or language difficulties
* Prior knee arthroplasty in the joint to operate
* Prior arthroplasty in another weight-bearing joint within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477
Dates: Start 2007-01; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Physical functioning as measured with the Western Ontario and McMasters osteoarthritis index

SECONDARY OUTCOMES:
Leg-specific pain and stiffness as measured with the WOMAC
The Lequesne Knee Score
The physical component summary of the SF-36
EuroQoL-5D
Patient satisfaction
Balance abilities as investigated with the Biodex Stability System®
Motoric coordination as assessed by a shortened version of the "Dortmunder modified Romberg Test for Seniors"
Proprioception assessed according to guidelines established by Barrack and Swanik
Axis relations evaluated by postoperative standardized lateral and AP X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Hassenpflug, Prof. Dr., Study Chair — University of Schleswig-Holstein, Kiel Medical Center; Thoralf R Liebs, Dr., Principal Investigator — University of Schleswig-Holstein, Kiel Medical Center
Locations (8):
- Germany (8):
  - University of Mannheim, Center for Orthopaedic Surgery and Traumatology, Mannheim, Baden-Wurttemberg
  - University of Regensburg, Department of Orthopaedic Surgery, Bad Abbach, Bavaria
  - University of Würzburg, Department of Orthopaedic Surgery, Würzburg, Bavaria
  - DIAKO Ev. Diakonie-Hospital gGmbH, Clinic for Orthopaedic Surgery and Traumatology, Bremen, City state Bremen
  - Schön-Klinikum Hamburg-Eilbek, Department of Orthopedic Surgery and Traumatology, Hamburg, Hamburg
  - University of Cologne, Department of Orthopaedic Surgery, Cologne, Northrhine-Westfalia
  - University of Schleswig-Holstein, Kiel Medical Center, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Center for Musculoskeletal Surgery, Berlin, State of Berlin